CLINICAL TRIAL: NCT01957423
Title: Immune Response Regulation and Nutritional Status of Crohn's Disease Patients Under Anti-TNF-alpha and Azathioprine Therapy.
Brief Title: Immune Response Regulation and Nutritional Status of the Crohn's Disease Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, PhD Maria Marluce dos Santos Vilela, MD, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 1099.0.146.000-11
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; whey protein; soy protein; nutritional status; activity of disease
MeSH Terms: conditions — Crohn Disease | interventions — Whey Proteins; Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whey protein (Experimental): Whey protein was provided as sachets with 15g. Patients were advised to consume two sachets per day (amounting to 22.4g of protein) mixed with food or a cold beverage, for 16 weeks. All patients remained on an unrestricted diet and did not receive nutritional advice.
  Interventions: Dietary Supplement: Whey protein
- Soy protein (Active Comparator): Soy protein was provided as sachets with 15g. Patients were advised to consume two sachets per day (amounting to 22.4g of protein) mixed with food or a cold beverage, for 16 weeks. All patients remained on an unrestricted diet and did not receive nutritional advice.
  Interventions: Dietary Supplement: Soy protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Whey protein was provided as sachets with 15g. Patients were advised to consume two sachets per day (amounting to 22.4g of protein) mixed with food or a cold beverage, for 16 weeks. All patients remained on an unrestricted diet and did not receive nutritional advice.
  Arms: Whey protein
Dietary Supplement: Soy protein — Soy protein was provided as sachets with 15g. Patients were advised to consume two sachets per day (amounting to 22.4g of protein) mixed with food or a cold beverage, for 16 weeks. All patients remained on an unrestricted diet and did not receive nutritional advice.
  Arms: Soy protein

SUMMARY:
The objective of this study was to evaluate the effect of Whey Protein (WP) and Soy Protein (SP) nutritional supplements on nutritional status and disease activity in Crohn's disease patients.

DETAILED DESCRIPTION:
The patients were split into two groups: one group was supplemented with whey protein and the other, with soy protein. Participants were assessed at three moments: before starting the intervention and after 8 and 16 weeks. The nutritional status and body composition were measured using bioimpedance analysis, anthropometry and albumin and pre-albumin dosages. Dietary intake was determined by 24-h dietary recalls. The disease activity was evaluated by Crohn's Disease Activity Index, serum cytokines and C-reactive protein dosages.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease patients treated with azathioprine or anti-tumor necrosis factor-alpha (anti-TNF-alpha) or azathioprine and anti-TNF-alpha

Exclusion Criteria:

* smokers
* who were using other medication or nutritional supplements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Body mass index | 16 weeks
  Body mass index (BMI) was calculated from weight and height (kilograms per meter squared) and classified according to the World Health Organization.

SECONDARY OUTCOMES:
Body fat percentage | 16 weeks
  Body fat was measured using bioimpedance analysis. Whole-body resistance and reactance were measured using a tetrapolar bioelectrical impedance analyzer in accordance with the manufacturer's guidelines (BIODYNAMICS, Model 310e).
Body lean percentage | 16 weeks
  The body lean mass was measured using bioimpedance analysis. Whole-body resistance and reactance were measured using a tetrapolar bioelectrical impedance analyzer in accordance with the manufacturer's guidelines (BIODYNAMICS, Model 310e).
Mid-arm circumference | 16 weeks
  Mid-arm circumference was obtained using the tape measure.
Mid-arm muscle circumference | 16 weeks
  Mid-arm muscle circumference was calculated from mid-arm circumference and triceps skin fold thickness.
Corrected arm muscle area | 16 weeks
  Corrected arm muscle area was calculated from mid-arm circumference and triceps skin fold thickness.
Crohn's Disease Activity Index | 16 weeks
  The Crohn's Disease Activity Index was used for evaluation of disease activity.
C-reactive protein | 16 weeks
Serum albumin | 16 weeks
Pre-albumin | 16 weeks
Triceps skin fold thickness | 16 weeks
  Triceps skin fold thickness was obtained using the Lange skin fold caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Maria MS Vilela, MD PhD, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil